CLINICAL TRIAL: NCT06042244
Title: Multimodal Exercise Training to Reduce Frailty in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00149742
Record Dates: First submitted 2023-07-21; First posted 2023-09-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Frailty
MeSH Terms: conditions — Multiple Sclerosis; Frailty | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Participants randomized to the control group will be put on a waitlist (passive control group) for 6 weeks. Upon completion of post-training assessment, participants in the control group will be able to receive the intervention, if they wish so.
  Interventions: Other: Waitlist
- Multimodal Exercise Group (Experimental): Participants will complete 15 minutes of virtual reality treadmill training (VRTT), followed by 30 minutes of progressive evidence-based resistance training (RT), followed by other 15 minutes of VRTT.
  Interventions: Other: Multimodal Exercise Group

INTERVENTIONS:
Other: Multimodal Exercise Group — Listed in arm/ group descriptions
  Arms: Multimodal Exercise Group
Other: Waitlist — listed in arm/group description
  Arms: Control Group

SUMMARY:
Study Significance: This proposed investigation is designed to examine the feasibility of an exercise-based intervention to reduce frailty in people living with MS. The proposed research will be the first to establish the feasibility of targeting frailty in pwMS and will begin to examine the dynamic nature of frailty in MS. These advances will pave the way for planned prospective studies toward effective targets for diagnostics, and rehabilitation of frailty in MS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged 40-65 years old to be enrolled in this study.
* Subjects must meet 3 of 5 frailty criteria (weight loss; exhaustion; weakness; slowness; inactivity) to be considered.
* Subjects must have a confirmed diagnosis of MS by the treating neurologist
* be free from MS relapses in the last 30 days
* have an Expanded Disability Status Scale (EDSS) score ≤ 6.0
* be fluent in spoken and written English.

Exclusion Criteria:

* unable to walk unassisted for at least ten meters
* are diagnosed with other clinically important neurological conditions (such as Parkinson's Disease, epilepsy, etc.)
* exhibit severe cognitive impairment (as determined by a Mini-Cog score <3)
* are diagnosed with active psychiatric problems.
* unstable cardiovascular conditions (e.g., malignant arrhythmias, critical mitral stenosis, clinically severe left ventricular outflow obstruction, critical proximal coronary artery stenosis)
* arthritis of the lower limbs
* acute lower back or lower limbs pain
* rheumatic and/or severe orthopedic problems that may interfere with resistance training.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 6 weeks
  Preliminary efficacy of multimodal exercise in improving frailty [Time frame: The EFIP outcome will be assessed at baseline and at 6-weeks post-intervention] Frailty will be evaluated through the Evaluative Frailty Index for Physical Activity (EFIP).

CONTACTS AND LOCATIONS:
Locations (1):
- Landon Center On Aging, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Zanotto T, Kumar DP, Tabatabaei A, Lynch SG, He J, Herda TJ, Devos H, Thiyagarajan R, Chaves L, Seldeen K, Troen BR, Sosnoff JJ. Multimodal exercise training to reduce frailty in people with multiple sclerosis: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2024 Apr 22;10(1):65. doi: 10.1186/s40814-024-01496-2. PMID 38650042